CLINICAL TRIAL: NCT07107126
Title: A Phase 1 Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Leukemia Activity of RPT1G in Patients With Acute Myeloid Leukemia (AML) and High-Risk Myelodysplastic Syndromes (MDS)
Brief Title: Safety and Proof-of-Concept Study of RPT1G in Adults With Acute Myeloid Leukemia and High-Risk Myelodysplastic Syndromes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Remedy Plan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RPT1G-1002
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Starting Dose of RPT1G
  Interventions: Drug: RPT1G
- Cohort 2 (Experimental): 2nd ascending dose of RPT1G
  Interventions: Drug: RPT1G
- Cohort 3 (Experimental): 3rd ascending dose of RPT1G
  Interventions: Drug: RPT1G

INTERVENTIONS:
Drug: RPT1G — RPT1G is a selective hyperbolic NAMPT inhibitor. RPT1G is administered orally.

SUMMARY:
The main goals of this study are to learn if RPT1G is safe and tolerable and to determine the best dose and schedule of RPT1G for patients with relapsed or refractory acute myeloid leukemia (AML) and high-risk myelodysplastic syndromes (MDS).

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Histological confirmation of AML (ELN 2022 criteria) that relapsed and/or refractory AML or high-risk MDS as defined by International Consortium for MDS (icMDS) 2023 criteria that have received appropriate standard of care therapy, in the opinion of the investigator or declined receipt of these
* Organ function/reserve as per the following laboratory criteria:
* Hepatic: Aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤2.5 x ULN, and total bilirubin <2 x ULN (except for study patients with known Gilbert's where 1.5 x UL of the subject's baseline or in the case of suspected Gilbert's syndrome where a maximum total bilirubin level of 4.0 mg/dL is acceptable) for the local laboratory. If due to disease, higher values may be approved after discussion with medical monitor.
* Renal: Adequate renal function as defined by calculated creatinine clearance >50 mL/min for the CLIA certified local laboratory. Creatinine clearance must be calculated by Cockcroft-Gault equation.

Key Exclusion Criteria:

* Patients without evidence of blood or marrow involvement
* Acute promyelocytic leukemia
* Symptomatic central nervous system involvement by AML
* Clinical signs/symptoms of leukostasis requiring urgent therapy
* Active infections
* Radiotherapy <14 days prior to the first day of RPT1G administration
* Ongoing complications from prior therapy
* Prior or concurrent malignancy
* Any other condition, therapy, treatment, or comorbidity that leads the investigator to determine that the study is not in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of RPT1G in patients with acute myeloid leukemia and high-risk myelodysplastic syndromes | 3 years
  Incidence of adverse events and serious adverse events and frequency of treatment-emergent adverse events leading to discontinuation of study treatment